CLINICAL TRIAL: NCT05591651
Title: The Effectiveness of Hyaluronic Acid for the Treatment of Damaged Nipples in Breastfeeding Women: a Double-blind Randomised, Controlled Trial
Brief Title: Hyaluronic Acid for the Treatment of Damaged Nipples in Breastfeeding Women
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Specijalisticka Pedijatrijska Ordinacija prim.mr.sc. Maja Stimac, Specijalist Pedijatrije Sspecijalnosti Neonatologije (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 123456
Record Dates: First submitted 2022-10-13; First posted 2022-10-24 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Cracked Nipple; Breastfeeding; Healing Wound
Keywords: hyaluronic acid; cracked nipple; breastfeeding
MeSH Terms: conditions — Breast Feeding | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Preparation with hyaluronic acid (Experimental): Treatment of damaged nipple skin: Preparation with hyaluronic acid. The hyaluronic acid preparation will contain white vaseline and 0.2% sodium hyaluronate in a 30 g container.
  Interventions: Drug: Treatment of damaged nipple skin: Preparation with hyaluronic acid
- Neutral Preparation without hyaluronic acid (Experimental): Treatment of damaged nipple skin: Neutral preparation without hyaluronic acid. The neutral preparation will contain white vaseline only, in a 30 g container, and wiil have the same appearance and fragrance as the active preparation.
  Interventions: Drug: Treatment of damaged nipple skin: Neutral preparation without hyaluronic acid

INTERVENTIONS:
Drug: Treatment of damaged nipple skin: Preparation with hyaluronic acid — The active preparation will be applied for five days, locally on the damaged nipple skin after every second breastfeeding session, and at least four times in 24 hours, alternating it with breast milk.
  Arms: Preparation with hyaluronic acid
Drug: Treatment of damaged nipple skin: Neutral preparation without hyaluronic acid — The neutral preparation, containing only white vaseline, will be applied for five days, locally on the damaged nipple skin after every second breastfeeding session, and at least four times in 24 hours, alternating it with breast milk.
  Arms: Neutral Preparation without hyaluronic acid

SUMMARY:
Previous studies have shown that application of hyaluronic acid preparations to wounds of the skin and mucosa have a beneficial effect.

There is a lack of studies showing the effect of applying hyaluronic acid preparations to treat damaged nipple skin in breastfeeding mothers.

This study aims to determine the effect of applying a hyaluronic acid preparation to damaged nipple skin in breastfeeding women.

DETAILED DESCRIPTION:
A randomised, controlled, parallel, double-blinded clinical trial will be performed in the Breastfeeding Support Unit of the Health Centre 'Dom zdravlja' in Osijek-Baranja County, Croatia, in 2022.

A randomised controlled study design has been chosen for this trial to compare two ways of treating damaged nipples in breastfeeding women. Participants will be randomly divided into two groups. The randomisation procedure will ensure the reliability of the results. Participants are breastfeeding mothers, with damaged nipples, and their newborn babies. Eligible mothers will be directed to the Breastfeeding Support Unit by the Health Centre's Health Visitors during regular home visits. Participants will be included in the study only if both mother and child meet the inclusion criteria.

Participants will be divided into two groups by simple randomisation: a group receiving a hyaluronic acid preparation and a control group receiving a placebo preparation. Allocation will be performed using a computer-generated list of random numbers. The allocator will know which participant receives which preparation, whereas the main researcher and the participants will not know which preparation is used by any participants. All pregnancy and birth data will be collected from the medical documentation of the mother and the child.

The preparation containing hyaluronic acid and the neutral agent will be prepared in the Galenska laboratory, Ljekarna Srce, Osijek-Baranja County. The hyaluronic acid preparation will contain white vaseline and 0.2% sodium hyaluronate in a 30 g container. The preparation will be applied for five days, locally on the nipple skin area after every second breastfeeding session and at least four times in 24 hours, alternating it with breast milk. The hyaluronic acid preparation will be distributed in the same packaging as the neutral agent used by the control group. The control group participants will apply the neutral agent containing only white vaseline for five days after every second breastfeeding session and at least four times in 24 hours, alternating it with breast milk. All mothers will be advised to wash the nipple skin with water before the next breastfeed.

The participants will be examined four times during their first postpartum month in the Breastfeeding Support Unit of the Health Centre 'Dom zdravlja'. The first check-up will occur 72 to 120 hours postpartum when the participants will be introduced to the study, provide consent for participation in the study, and, according to the allocator's instructions, will receive the preparation to treat the damaged nipple skin. Then, the researcher will advise the participants on how to position their babies during breastfeeding and correct possible irregularities.

The next check-up will occur at the Breastfeeding Support Unit on the seventh postpartum day when the condition of the damaged skin will be evaluated. The other check-ups will occur on the 10th and 30th postpartum days in the Breastfeeding Support Unit. During every checkup, the condition of the damaged nipple skin will be evaluated, participants will estimate the soreness on a visual analogue scale, and the mother's satisfaction with the treatment method will be assessed. During every visit, the baby's diet will be checked and noted, and possible side effects in the mother and child will be recorded.

Nipple healing will be measured using the Nipple Trauma Score (NTS), and the measurement will be done by the lead researcher. During the nipple skin checkup, the following NTS interpretation will be applied: 0) no macroscopically visible skin changes; 1) erythema or edema or combination of both; 2) superficial damage with or without scab formation of less than 25% of the nipple surface; 3) superficial damage with or without scab formation of more than 25% of the nipple surface; 4) partial-thickness wound with or without scab formation of less than 25% of the nipple surface; 5) partial-thickness wound with or without scab formation of more than 25% of the nipple surface.

Nipple pain will be estimated using an adapted visual analogue scale (VAS). The pain scale is marked by numbers 0 to 10, where 0 means no pain, and 10 is the highest pain imaginable. The mother will decide on the VAS scale, which measure best fits her pain: 0) no pain, feeling that the child is moving my breast; 1-2) minimal discomfort and pain; 3-5) moderate pain; 6-8) severe pain; 9-10) the severest pain I can imagine.

The mother's satisfaction with the applied preparation will be measured using a Likert scale. The mother will choose one of the given answers: 1- Very dissatisfied; 2 - Dissatisfied; 3 - Neutral/ don't have an opinion; 4 - Satisfied; and 5 - Very satisfied.

During Breastfeeding Support Unit visits, mothers will be asked whether they have noticed any side effects in either themselves or their child. In addition, infant feeding will be monitored, specifically if breastfeeding is exclusive during the first month. World Health Organisation (WHO) definitions will be used, according to which exclusive breastfeeding is defined as feeding the child with breast milk only, without any other fluids or food, besides minerals and vitamins.

The researcher aims to find the middle effect in the difference of numerical variables between the participants in the two independent groups, with a 0.05 level of significance and 0.08 statistical power; hence, the minimal sample needed is 64 participants per group or 128 participants in total. Assuming a 20% loss of participation within the study group, the expected sample is 160 participants to detect a statistically significant difference.

This study will use rigorous scientific procedures to investigate whether hyaluronic acid is more efficient in treating nipple skin damage in breastfeeding mothers than a neutral agent. If the intervention proves to be effective, i.e. if there is faster healing of the damaged nipple skin and a reduction in pain, it may be a potential way of easing breastfeeding difficulties of mothers at the beginning of the breastfeeding period, which might lead to a more significant percentage of breastfed children which will benefit the whole of society.

ELIGIBILITY:
Inclusion Criteria:

* for mothers: a breastfeeding mother, living or residing in Osijek, with nipple skin damage (NTS 1, 2, 3, 4, or 5).
* for babies: newborns from a singleton pregnancy, of gestational age from 37 to 42 weeks, with a birth weight of 2,500 to 4,500 grams.

Exclusion Criteria:

* for mothers: mothers who do not breastfeed, mothers not living or residing in Osijek, mothers without nipple skin damage and mothers using other preparations for healing sore nipples (shells, pads).
* for children: visible anomalies in the newborn which may affect the breastfeeding process, newborns that required admission to the neonatal unit

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Healing of damaged nipples | 30 days
  Nipple healing will be measured using the Nipple Trauma Score (NTS). Measurements will be performed by the lead researcher using the following scale: 0) no macroscopically visible skin changes; 1) erythema or edema or combination of both; 2) superficial damage with or without scab formation of less than 25% of the nipple surface; 3) superficial damage with or without scab formation of more than 25% of the nipple surface; 4) partial-thickness wound with or without scab formation of less than 25% of the nipple surface; 5) partial-thickness wound with or without scab formation of more than 25% of the nipple surface.
Level of nipple pain | 30 days
  Nipple pain will be estimated using an adapted VAS.The pain scale is marked by numbers 0 to 10, where 0 means no pain, and 10 is the highest pain imaginable. The mother will decide on the VAS scale, which measure best fits her pain: 0) no pain, feeling that the child is moving my breast; 1-2) minimal discomfort and pain; 3-5) moderate pain; 6-8) severe pain; 9-10) the severest pain I can imagine.

SECONDARY OUTCOMES:
Mother's satisfaction with allocated treatment | 30 days
  The mother's satisfaction with the applied preparation will be measured using a Likert scale. The mother will be able to choose one of the following options: 1- Very dissatisfied; 2 - Dissatisfied; 3 - Neutral/ don't have an opinion; 4 - Satisfied; and 5 - Very satisfied.
Exclusive breastfeeding rates at days 3, 7, 10, and 30 postpartum. | 30 days
  During the Breastfeeding Support Unit visits, mothers wiil be asked by the lead researcher how their newborn was fed in the previous 24h, and since the last visit. WHO breastfeeding definitions wiil be used, according to which exclusive breastfeeding is defined as receiving only human milk, without any other fluids or food, apart from minerals and vitamins.
Side effects in mother and child | 30 days
  During Breastfeeding Support Unit visits, mothers will be asked whether they have noticed any side effects on themselves or on their infants.

CONTACTS AND LOCATIONS:
Overall Officials: Maja Štimac, MD; Mr.sc., Principal Investigator — Specijalistička pedijatrijska ordinacija prim.mr.sc.Maja Štimac
Locations (1):
- Savjetovalište za dojenje, Dom zdravlja Osječko-baranjske županije, Osijek, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tait P. Nipple pain in breastfeeding women: causes, treatment, and prevention strategies. J Midwifery Womens Health. 2000 May-Jun;45(3):212-5. doi: 10.1016/s1526-9523(00)00011-8. PMID 10907330
- [Background] Abou-Dakn M, Fluhr JW, Gensch M, Wockel A. Positive effect of HPA lanolin versus expressed breastmilk on painful and damaged nipples during lactation. Skin Pharmacol Physiol. 2011;24(1):27-35. doi: 10.1159/000318228. Epub 2010 Aug 18. PMID 20720454
- [Background] Shaharudin A, Aziz Z. Effectiveness of hyaluronic acid and its derivatives on chronic wounds: a systematic review. J Wound Care. 2016 Oct 2;25(10):585-592. doi: 10.12968/jowc.2016.25.10.585. PMID 27681589
- [Background] Torretta S, Marchisio P, Rinaldi V, Carioli D, Nazzari E, Pignataro L. Endoscopic and clinical benefits of hyaluronic acid in children with chronic adenoiditis and middle ear disease. Eur Arch Otorhinolaryngol. 2017 Mar;274(3):1423-1429. doi: 10.1007/s00405-016-4327-4. Epub 2016 Oct 1. PMID 27695944